# Examining the Efficacy of a Tri-Compartment Unloader Knee Brace During Physical Rehabilitation in Non-Surgical Patients with Anterior Knee Pain

Study Protocol

NCT05428332

June 28, 2022

# Study: Examining the Efficacy of a Tri-Compartment Unloader Knee Brace during Physical Rehabilitation in Non-Surgical Patients with Anterior Knee Pain

- Brief Summary: This study will examine clinical outcomes related to pain and function in patients with anterior knee pain (i.e. focal patella and/or trochlea cartilage defect(s), patellofemoral arthritis) before and after standard of care, non-surgical management with and without the addition of a Tri-Compartment Unloader (TCU) knee brace during activities of daily living. Randomly selected participants will wear a TCU brace for several weeks during physical therapy and activities of daily living that is designed to reduce compressive forces in all three compartments of the knee during weight-bearing flexion. Our hypothesis is that TCU bracing will improve clinical outcomes related to pain and function.
- The standard of care will be the same for all patients and will include NSAIDs, tylenol,
   PT at Stanford, counselling regarding weight optimization.
- Injection therapy for knee osteoarthritis will not be performed during the study period.
   Patients will be excluded if they have had an injection within 3 months of study enrollment.
- Patients with major mechanical symptoms or those otherwise considered surgical candidates will be excluded from this study during initial evaluation.
- The length and follow up schedule will be the same for all patients.
- The only difference in groups will be the presence or absence of TCU brace usage.

#### **Study Design**

 Participants: Non-surgical patients with patellofemoral defects and chronic patellofemoral knee pain

• Sample size: 20 participants (10 per group)

#### **Study Groups:**

| Group | Interventions/ Treatments |
|---|---|
| Experimental:<br>TCU bracing | <ul> <li>Device: TCU Knee Brace (Levitation 2)</li> <li>Participants will be instructed to wear a TCU knee brace for a minimum of 3 hours per day during activities of daily living and undergo Dr. Sherman's standard of care rehabilitation protocol.</li> <li>Participants will use the TCU knee brace during PT exercises, as determined by the PT team</li> <li>Participants will undergo Dr. Sherman's standard of care rehabilitation protocol, including NSAIDs, tylenol, PT.</li> </ul> |
| Control: | No Device - Participants will undergo Dr. Sherman's standard of care rehabilitation protocol only. |

**Outcomes Measures** Outcomes will be measured at baseline (before any intervention), 6 weeks after commencing rehabilitation, and 3 months after commencing rehabilitation.

## **Primary Outcome Measures:**

- 1. Knee Injury and Osteoarthritis Outcome Score (KOOS)
- 2. Pain intensity during activities of daily living (including walking, going up and down stairs, squatting, and sit to stand) measured with a Visual Analog Scale (VAS)

## **Secondary Outcome Measures:**

- 3. Quality of life (EQ-5D)
- 4. Physical activity levels (Lower Extremity Activity Scale/LEAS)
- 5. Quadricep strength (girth)
- 6. Effusion grade
- 7. Painful crepitus with deep knee flexion
- 8. Knee range of motion
- 9. PET-MRI at baseline, 3 months and 6 months per Feliks Kogan protocol

#### **Inclusion Criteria:**

- 1. Anterior knee pain that worsens when the knee is flexed and bearing weight
- Patellofemoral chondral defect(s) or patellofemoral arthritis detected with standard of care x-ray and/or MRI
- 3. Kellgren and Lawrence grade 0-3 of PF joint
- 4. Able to wear the TCU knee brace for a minimum of 3 hours per day
- 5. Over 18 years old, can understand written English
- 6. Coronal knee alignment within 7 degrees of neutral
- 7. Must be able to fit within an off-the-shelf knee brace size provided by Company
- 8. Must be able to participate in rehabilitation through Stanford

#### **Exclusion Criteria:**

- 1. Surgical intervention definitely indicated (major mechanical symptoms/failed substantial previous conservative measures) on the affected knee within the next year
- 2. Use of another brace designed to unload the knee or manage knee pain during the study
- 3. Varus/Valgus joint alignment > 7 degrees
- 4. Inability to be fit properly in an off-the-shelf brace provided by the Company
- 5. BMI >40
- 6. Bilateral knee symptoms